CLINICAL TRIAL: NCT06016595
Title: Retrospective Data Analysis in Chronic Prostatitis/Chronic Pelvic Pain Syndrome Patients: Evaluation of the Relationship Between Presence of Microorganism and Severity of Symptom
Brief Title: Chronic Prostatitis/Chronic Pelvic Pain Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Ass. Prof., Hisar Intercontinental Hospital
Other Study IDs: 16.08.2023/23-43
Record Dates: First submitted 2023-08-16; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Prostatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- singel
  Interventions: Diagnostic Test: Chronic prostatitis/chronic pelvic pain syndrome

INTERVENTIONS:
Diagnostic Test: Chronic prostatitis/chronic pelvic pain syndrome — Chronic prostatitis/chronic pelvic pain syndrome UPOINT

SUMMARY:
Chronic prostatitis/chronic pelvic pain syndrome (CPPS) is a common health problem among men and can cause severe quality of life. The pathophysiology of CPPS is still poorly understood and effective treatments are a challenging issue. This study aims to investigate the possible relationship between the presence of microorganisms in the prostatic fluid and symptom severity by presenting a retrospective analysis based on data from CPPS patients.

DETAILED DESCRIPTION:
This study is based on data from 112 CPPS patients aged 20-60 years. Various variables such as demographic information of the patients, International Prostate Symptom Score (I-PSS), which evaluates CPPS symptoms, inflammatory and non-inflammatory symptoms of CPPS, baseline scores of the International Index of Erectile Function (IIEF), which evaluates erectile function, and the presence of microorganisms in the prostate fluid were analyzed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with chronic prostatitis/chronic pelvic pain syndrome and whose prostate fluid was taken with prostate massage and androflor testis were studied were included.

Exclusion Criteria:

* acute and/or chronic bacterial prostatitis, active history of genitourinary cancer, history of recent prostate surgery the diagnosis of neurological diseases affecting the bladder was determined

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients with chronic prostatitis were included in the study.
Study Population: This study is based on data from 112 CPPS patients aged 20-60 years. Various variables such as demographic information of the patients, International Prostate Symptom Score (I-PSS), which evaluates CPPS symptoms, inflammatory and non-inflammatory symptoms of CPPS, baseline scores of the International Index of Erectile Function (IIEF), which evaluates erectile function, and the presence of microorganisms in the prostate fluid were analyzed retrospectively.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Correlation between androflor pcr positive patients and uopint and nih-cpsi | 2 years
  Those with positive and negative Androflor PCR test will be evaluated. testicular torsion

CONTACTS AND LOCATIONS:
Locations (1):
- Hisar Intercontinental Hospital, Istanbul, Turkey (Türkiye)